CLINICAL TRIAL: NCT07405801
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Inavolisib Plus Ribociclib Plus Fulvestrant Versus Placebo Plus Ribociclib Plus Fulvestrant in Patients With Endocrine- Resistant Hormone-Receptor-Positive, HER2-Negative Advanced Breast Cancer With Chromosome 8P Loss and Without a PIK3CA Mutation
Brief Title: A Phase II Study Evaluating the Efficacy and Safety of Inavolisib Plus Ribociclib Plus Fulvestrant Versus Placebo Plus Ribociclib Plus Fulvestrant in Participants With Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO46274; 2025-523013-28-00 (EU CTIS Number)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; ribociclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inavolisib + Ribociclib + Fulvestrant (Experimental): Participants will receive inavolisib, ribociclib and fulvestrant.
  Interventions: Drug: Inavolisib; Drug: Ribociclib; Drug: Fulvestrant
- Placebo + Ribociclib + Fulvestrant (Placebo Comparator): Participants will receive placebo, ribociclib and fulvestrant.
  Interventions: Drug: Ribociclib; Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Inavolisib — Inavolisib will be administered as per the schedule mentioned in the protocol.
  Arms: Inavolisib + Ribociclib + Fulvestrant
Drug: Ribociclib — Ribociclib will be administered as per the schedule mentioned in the protocol.
Drug: Fulvestrant — Fulvestrant will be administered as per the schedule mentioned in the protocol.
Drug: Placebo — Placebo will be administered as per the schedule mentioned in the protocol.
  Arms: Placebo + Ribociclib + Fulvestrant

SUMMARY:
A study to evaluate the efficacy and safety of triplet combination of inavolisib plus ribociclib and fulvestrant versus placebo plus ribociclib and fulvestrant in the first-line setting in participants with endocrine-therapy-resistant hormone receptor (HR)-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) advanced breast cancer (ABC) with chromosome 8p loss (chr8p loss) and without PIK3CA mutation.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with histologically or cytologically confirmed carcinoma of the breast that is locally advanced or metastatic and is not amenable to surgical or radiation therapy with curative intent
* Documented estrogen receptor (ER)-positive and/or progesterone receptor (PR)-positive tumor according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines, defined as >=1% of tumor cells stained positive based on the most recent tumor biopsy and assessed locally (Allison et al. 2020)
* Participants must not have received any prior systemic therapy for locally advanced unresectable or metastatic breast cancer (mBC) and must have progressed during adjuvant endocrine-based treatment or within 12 months after completing adjuvant endocrine-based therapy with an aromatase inhibitor or tamoxifen
* Confirmed biomarker eligibility as documented through central laboratory testing of a tumor tissue sample documenting both the lack of a phosphatidylinositol-4,5-biphosphate 3-kinase catalytic subunit alpha gene (PIK3CA) mutation and the presence of heterozygous loss of chromosome 8p (i.e., PIK3CAnmd and chr8p loss)
* Measurable disease per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)

Exclusion Criteria:

* Metaplastic breast cancer
* Radiotherapy within 2 weeks before randomization
* Appropriate for treatment with cytotoxic chemotherapy at time of entry into the study, as per national or local treatment guidelines (e.g., participants with visceral crisis)
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Known and untreated, or active Central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Participants with a history of treated CNS metastases are eligible
* Any history of leptomeningeal disease or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-12-19 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Confirmed Objective Response (cORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Percentage of Participants with Clinical Benefit (CBR) | Up to approximately 2 years
Percentage of Participants with Adverse Events (AEs) | Up to approximately 2 years
Number of Participants Reporting Presence, Frequency, Severity, and/or Degree of Interference With Daily Function of Symptomatic Treatment Toxicities Assessed by NCI Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 2 years
Number of Participants Reporting Each Response Option for Treatment Side-effect Bother Single-item General Population, Question 5 (GP5) From the Functional Assessment of Cancer Therapy-General Questionnaire; (FACT-G) | Up to approximately 2 years
Change From Baseline in Symptomatic Treatment Toxicities as Assessed Through use of the PRO-CTCAE | Baseline, Up to approximately 2 years
Change from Baseline in Treatment Side-effect Bother as Assessed Through use of the FACT-G GP5 Item | Baseline, Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing